CLINICAL TRIAL: NCT03098966
Title: Evaluation of Trials of Labor After Previous Cesarean Section in Ain Shams University Maternity Hospital
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rehab Mohamed Abdelrahman, Lecturer of Obstetrics and Gynaecology Faculty of Medicine, Ain Shams University, Ain Shams University
Other Study IDs: TOLAC
Record Dates: First submitted 2017-03-28; First posted 2017-04-04 (Actual); Results first posted 2018-01-26 (Actual); Last update posted 2018-01-26 (Actual); Status verified 2017-06

CONDITIONS: Vaginal Birth After Cesarean

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study to evaluate the practice and short term maternal and perinatal outcomes of trial of labor after cesarean section offered to women at Ain Shams University Maternity Hospital (ASUMH) during the 3-year period from January 2013 to December 2015.

DETAILED DESCRIPTION:
This is a retrospective study that was performed at Ain Shams University Maternity Hospital.

The following data will be gathered (whenever available), tabulated and subjected to the proper statistical analysis:

History:

* Age
* Duration of marriage
* Inter-pregnancy interval
* Gestational age (by menstrual dates or US)
* Obstetric history (parity, mode of delivery, assisted vaginal delivery, previous vaginal birth after cesarean section, neonatal outcome)
* Present and past history of any medical, surgical or obstetric problems; history of infection after previous CS

General examination:

* General condition
* Vital data

Abdominal examination:

* Fundal level
* Estimated fetal weight (clinically or by US)
* Scar tenderness

Vaginal examination on admission:

* Cervical status
* Station of presenting part
* Membranes status
* Pelvic adequacy

Investigations performed:

* Complete Blood Count
* Ultrasonography

Intrapartum management:

* Progress and duration of labor according to partogram (or admission-delivery time)
* Intrapartum complications; placental abruption, uterine rupture, hysterectomy, complications during surgical intervention if any

Mode of delivery:

* Vaginal delivery (spontaneous, assisted, complications)
* Cesarean section (indication, scar dehiscence)

Postpartum Data:

* Postpartum hemorrhage
* Blood transfusion
* Neonatal outcome; fetal weight, birth trauma, Neonatal Intensive Care Unit admission, mortality

ELIGIBILITY:
Inclusion Criteria:

* Women admitted in labour
* One prior caesarean section
* Singleton pregnancy
* Vertex-presenting fetus

Exclusion Criteria:

* Prior high-risk uterine scar; uterine rupture, classical CS, hysterotomy or myomectomy
* Short inter-delivery interval (<12 months)
* Complications in the previous CS (e.g. puerperal sepsis)
* Obstetric indication for CS (either elective or emergency):

  * Placenta praevia
  * Placental abruption
  * Documented evidence of cephalopelvic disproportion
  * Fetal macrosomia (estimated fetal weight >4 kg)
  * Fetal anomalies interfering with vaginal delivery e.g. hydrocephalus
  * Fetal distress or non-reassuring Cardiotocography pattern

Ages: 20 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: This is a retrospective study that was performed at Ain Shams University Maternity Hospital Records of hospital admissions during the planned time frame were reviewed. Subjects eligible for conduction of a Trial Of Labor After Cesarean section (TOLAC), were included, while those ineligible for TOLAC were excluded from the study dataset.
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a retrospective study that was performed at Ain Shams University Maternity Hospital during the 3-year period from January 2013 to December 2015.
Groups:
- Trial Of Labour After Caesarean Section: The following data was gathered (whenever available), tabulated and subjected to the proper statistical analysis:
  -Vaginal examination on admission: Cervical status Station of presenting part Membranes status Pelvic adequacy
  -Intrapartum management: Progress and duration of labor according to partogram (or admission-delivery time) Intrapartum complications; placental abruption, uterine rupture, hysterectomy, complications during surgical intervention if any
  -Mode of delivery: Vaginal delivery (spontaneous, assisted, complications) Cesarean section (indication, scar dehiscence)
  -Postpartum Data: Postpartum hemorrhage Blood transfusion Neonatal outcome; fetal weight, birth trauma, Neonatal Intensive Care Unit admission, mortality
Period: Overall Study
Arm/Group | Trial Of Labour After Caesarean Section
Started | 368
Completed | 368
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Trial Of Labour After Caesarean Section
Number analyzed (Participants) | 368
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 368
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.6 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 368
  Male | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Egypt | 368

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Successful Vaginal Birth
Description: Mode of delivery: either successful vaginal birth after cesarean section or failed trial of labor (ending in emergency intrapartum cesarean section).
Time Frame: 24 hours after onset of trial of labor
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Of Labour After Caesarean Section
Number analyzed (Participants) | 368
Participants | 317

2. Secondary Outcome: Number of Participants Who Had Maternal Morbidity
Description: • Maternal morbidity:
  * Uterine rupture
  * Surgical injuries (during emergency CS)
  * Hemorrhage and blood transfusion
  * Peripartum hysterectomy
Time Frame: 48 hours after onset of trial of labor
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Of Labour After Caesarean Section
Number analyzed (Participants) | 368
Participants | 338

3. Secondary Outcome: Adverse Perinatal Outcomes
Description: • Adverse perinatal outcomes:
  * Apgar score
  * Neonatal Intensive Care Unit admission
  * Respiratory morbidity, e.g. transient tachypnoea of the newborn
  * Hypoxic ischaemic encephalopathy
  * Birth trauma
  * Mortality
Time Frame: 48 hours postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Trial Of Labour After Caesarean Section
Number analyzed (Participants) | 368
Participants | 332

ADVERSE EVENTS:
Time Frame: 1 month
Description: Trials of Labor After Previous Cesarean Section was performed and Adverse Events were assessed.
Arm/Group | Trial Of Labour After Caesarean Section
Serious Adverse Events (participants affected / at risk) | 0/368
Other Adverse Events (participants affected / at risk) | 0/368

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No